CLINICAL TRIAL: NCT01618422
Title: A Randomized, Parallel, Controlled Study to Evaluate the Role of Directly Observed Therapy Short Course-Plus (DOTS-Plus) Versus DOTS for Retreatment of Relapsed Pulmonary TB in Guangzhou.
Brief Title: Directly Observed Therapy Short Course-Plus Versus DOTS for Retreatment of Relapsed Pulmonary Tuberculosis in Guangzhou
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Prof David Shu Cheong Hui, Professor of Respiratory Medicine, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2008.286-T
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-11

CONDITIONS: Pulmonary Tuberculosis
Keywords: DOTS plus; DOTS; multidrug resistant tuberculosis (MDR TB)
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Directly Observed Therapy (DOTS) (Sham Comparator): The DOTS strategy (current standard strategy) consists of the following measures: political commitment, case detection through bacteriologic evaluation, standardized treatment with supervision and patient support, an effective drug supply system, and a reporting and recording system that allows assessment of treatment. The standard regimen for treatment of new cases of pulmonary TB consists of 6 months treatment, with 4 drugs in the initial phase including isoniazid, rifampicin, pyrazinamide, and either ethambutol or streptomycin, followed by two drugs in the continuation phase including isoniazid and rifampicin. In the treatment of previously treated cases, a standard regimen consisting of 8 months treatment will be used.
  Interventions: Other: Directly Observed Therapy (DOTS)
- Directly Observed Therapy (DOTS) plus (Active Comparator): The DOTS-Plus strategy (the strategy to be tested) includes additional measures including continuous drug resistance surveillance, culture, drug susceptibility testing for TB patients, and tailoring of individual drug regimen through the use of first and second-line drugs.
  Interventions: Other: Directly Observed Therapy (DOTS) plus

INTERVENTIONS:
Other: Directly Observed Therapy (DOTS) plus — The regimen used to treat MDR-TB comprises 5 to 6 drugs to which the organism is or likely to be susceptible for the initial 6 months, and then 3 to 4 drugs subsequently. In addition, TB cases with rifampicin resistance but not amounting to MDR-TB are also at risk of unfavourable treatment outcomes. The availability of pretreatment susceptibility test results will provide a guide in selection of drugs in treating such cases.
  Arms: Directly Observed Therapy (DOTS) plus
Other: Directly Observed Therapy (DOTS) — The DOTS strategy (current strategy) consists of the following measures: political commitment, case detection through bacteriologic evaluation, standardized treatment with supervision and patient support, an effective drug supply system, and a reporting and recording system that allows assessment of treatment. The standard regimen for treatment of new cases of pulmonary TB consists of 6 months treatment, with 4 drugs in the initial phase including isoniazid, rifampicin, pyrazinamide, and either ethambutol or streptomycin, followed by two drugs in the continuation phase including isoniazid and rifampicin. In the treatment of previously treated cases, a standard regimen consisting of 8 months treatment will be used.
  Arms: Directly Observed Therapy (DOTS)

SUMMARY:
This is a prospective, randomized, parallel, controlled study comparing the efficacy and outcomes in the retreatment of pulmonary Tuberculosis (TB) in Guangzhou in a group using pretreatment susceptibility tests in selection of chemotherapy regimens and that in another group without using pretreatment susceptibility test results. The investigators hypothesize that selecting drug treatment on the basis of known susceptibility tests would lead to improved outcome compared with empiric treatment.

DETAILED DESCRIPTION:
The aims are:1) To evaluate the efficacy and outcomes in the retreatment of pulmonary TB in Guangzhou by the use of pretreatment susceptibility tests in selection of chemotherapy regimens & 2) To study the predictive factors of unfavourable outcomes in the retreatment of pulmonary TB in Guangzhou, where unfavourable outcomes include treatment failures and relapses.

The patients will be randomized into either a) The DOTS strategy consisting of the following measures: political commitment, case detection through bacteriologic evaluation, standardized treatment with supervision and patient support, an effective drug supply system, and a reporting and recording system that allows assessment of treatment; or b) The DOTS-Plus strategy includes additional measures including continuous drug resistance surveillance, culture, drug susceptibility testing for TB patients, and tailoring of individual drug regimen through the use of first and second-line drugs.

The Primary end point is the 18-month combined treatment failure/ relapse (unfavourable outcome) among rifampicin resistant group. Secondary endpoints include the 30-month combined treatment failure/ relapse (unfavourable outcome) among rifampicin resistant group, multidrug resistant tuberculosis (MDR-TB) cases and all retreatment cases; Sputum smear/conversion rate at 2m, 3m, 8m, 12m, 18m, and 24m; Drug resistance rates to various drugs in particular rifampicin, and rate of MDR-TB. The predictive factors of unfavourable treatment outcomes (including failure and relapse) will be analysed.

The management of retreatment cases by DOTS alone is often problematic, especially when there is resistance to rifampicin, and treatment failure / relapse with further resistances might result. With implementation of the "DOTS-plus" strategy, Hong Kong (HK) has achieved a low MDR-TB prevalence of around 1%. This study will provide important data on the predictors of treatment failure/ relapse of retreatment cases and whether the DOTS-plus strategy can effectively reduce the failure/relapse rate and the prevalence rate of MDR-TB in Guangzhou. The project will provide useful data on the surveillance, epidemiology and public health control of TB with a regional (cross-border) significance.

ELIGIBILITY:
Inclusion Criteria:

All consecutive smear positive pulmonary TB patients aged at least 18 years, with past history of TB treatment, diagnosed with a new episode of active pulmonary TB requiring treatment will be recruited and randomized into two groups, with Group A with management based essentially on the DOTS strategy, while Group B based essentially on the DOTS-plus strategy.

Exclusion Criteria:

* Age < 18 yrs;
* New TB cases (without past history of anti-TB treatment) will be excluded because they have a much lower risk for MDR-TB than the retreatment cases.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2009-03; Primary Completion 2013-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Hui, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Guangzhou Chest Hospital, Guangzhou, Guangdong, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All consecutive patients suffering from tuberculosis (TB) of aged 18 years or older with past history of TB treatment of at least 1 month within 5 years and diagnosed with a new episode of sputum smear-positive pulmonary TB requiring treatment were recruited after informed consent.
Pre-assignment Details: Altogether 391 patients were assessed and after excluding those who did not meet inclusion criteria or refused to participate in the study, 225 patients were successfully randomized into DOTS (n=114) and DOTS plus (n=111).
Groups:
- DOTS Strategy: The standard regimen for treatment of new cases of pulmonary TB consists of 6 months treatment, with 4 drugs in the initial phase including isoniazid, rifampicin, pyrazinamide, and either ethambutol or streptomycin, followed by two drugs in the continuation phase including isoniazid and rifampicin. In the treatment of previously treated cases, a standard regimen consisting of 8 months treatment will be used.
- DOTS Plus: The DOTS-Plus strategy (the strategy to be tested) includes additional measures including continuous drug resistance surveillance, culture, drug susceptibility testing for TB patients, and tailoring of individual drug regimen through the use of first and second-line drugs. The regimen used to treat MDR-TB comprises 5 to 6 drugs to which the organism is or likely to be susceptible for the initial 6 months, and then 3 to 4 drugs subsequently. In addition, TB cases with rifampicin resistance but not amounting to MDR-TB are also at risk of unfavourable treatment outcomes. The availability of pretreatment susceptibility test results will provide a guide in selection of drugs in treating such cases.
  Directly Observed Therapy (DOTS) plus: The DOTS-Plus strategy (the strategy to be tested) includes additional measures including continuous drug resistance surveillance, culture, drug susceptibility testing for TB patients, and tailoring of individual drug regimen through the use of first and
Period: Overall Study
Arm/Group | DOTS Strategy | DOTS Plus
Started | 114 | 111
Completed | 114 | 111
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DOTS Strategy: The standard regimen for treatment of new cases of pulmonary TB consists of 6 months treatment, with 4 drugs in the initial phase including isoniazid, rifampicin, pyrazinamide, and either ethambutol or streptomycin, followed by two drugs in the continuation phase including isoniazid and rifampicin.
- DOTS Plus: Directly Observed Therapy (DOTS) plus: The DOTS-Plus strategy (the strategy to be tested) includes additional measures including continuous drug resistance surveillance, culture, drug susceptibility testing for TB patients, and tailoring of individual drug regimen through the use of first and second-line drugs. The regimen used to treat MDR-TB comprises 5 to 6 drugs to which the organism is or likely to be susceptible for the initial 6 months, and then 3 to 4 drugs subsequently. In addition, TB cases with rifampicin resistance but not amounting to MDR-TB are also at risk of unfavourable treatment outcomes. The availability of pretreatment susceptibility test results will provide a guide in selection of drugs in treating such cases.
- Total: Total of all reporting groups
Arm/Group | DOTS Strategy | DOTS Plus | Total
Number analyzed (Participants) | 114 | 111 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.25 (14.5) | 48.83 (17.07) | 48.05 (15.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 86 | 84 | 170
X ray lesions severity [Number; unit: participants] — Severity of chest x-ray (CXR) lesions is graded as follows:
  Mild: total area of involvement involving less than the size of right upper lobe; Moderate: total area of involvement was less than the size of right lung field but equal or bigger than right upper lobe; Severe: total area of involvement was bigger than right lung field.
  participants
    Mild | 34 | 18 | 52
    Moderate | 45 | 47 | 92
    Severe | 35 | 46 | 81
X ray showing cavitation [Number; unit: participants]
  Positive | 54 | 59 | 113
  Negative | 60 | 52 | 112
Sputum tuberculosis culture [Number; unit: participants]
  not available | 23 | 21 | 44
  Culture grew Mycobacterium tuberculosis complex | 79 | 77 | 156
  Culture grew non-tuberculosis mycobacterium | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Suffering From Treatment Failure/ Relapse (Unfavourable Outcome) Among Rifampicin Resistant Group.
Description: Cure (Completed for 8 months or more of therapy and culture converted in the last month of treatment, and on at least one previous occasion; for multidrug resistant TB (MDR-TB) switched to definitive second line therapy per protocol in the DOTS-plus group, sustained culture conversion for at least 6 months after initiation of second line therapy and no evidence of culture reversion up to the scheduled follow-up point); Treatment failure: not culture converted at 5 months or later; Defaulted: having interrupted treatment for 2 consecutive months or more; Transfer out: having been transferred to another recording and reporting unit and for whom the treatment outcome is not known; Death: a patient who died for any reason during the course of treatment Diagnosis revised: diagnosis revised to non-tuberculous mycobacterial infection or colonisation.
  Withdrawal: physician-initiated withdrawal for adverse effects, protocol violation or patient's decision to withdraw.
Time Frame: 18-month
Measure: Number; unit: participants
Arm/Group | DOTS Strategy | DOTS Plus
Number analyzed (Participants) | 114 | 111
participants
  Number of participants with treatment failure | 12 | 8
  Number of participants with cure | 67 | 73
  Number of participants with treatment completion | 0 | 0
  Number of participants defaulted follow up visit | 0 | 2
  Number of participants who were transferred out | 12 | 10
  Number of participants who were still on treatment | 2 | 0
  Number of death | 2 | 2
  Number of participants with diagnosis revised | 12 | 13
  Number of participants who withdrew from the study | 7 | 3

ADVERSE EVENTS:
Time Frame: 18 months
Groups:
- DOTS Strategy: The DOTS strategy (current strategy) consists of the following measures: political commitment, case detection through bacteriologic evaluation, standardized treatment with supervision and patient support, an effective drug supply system, and a reporting and recording system that allows assessment of treatment. The standard regimen for treatment of new cases of pulmonary TB consists of 6 months treatment, with 4 drugs in the initial phase including isoniazid, rifampicin, pyrazinamide, and either ethambutol or streptomycin, followed by two drugs in the continuation phase including isoniazid and rifampicin (2HRZE/4HR or 2HRZS/4HR). In the treatment of previously treated cases, a standard regimen consisting of 8 months treatment will be used (2HRZES/1HRZE/5HRE).
Arm/Group | DOTS Strategy | DOTS Plus
Serious Adverse Events (participants affected / at risk) | 2/114 | 2/111
Other Adverse Events (participants affected / at risk) | 0/114 | 0/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOTS Strategy (N=114) | DOTS Plus (N=111)
Death (Infections and infestations) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No